CLINICAL TRIAL: NCT01304979
Title: 'Acupuncture Therapy' for Pain and Function Recovery in Spine Surgery Patients
Acronym: Acuspine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 035-10
Record Dates: First submitted 2010-10-22; First posted 2011-02-28 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Pain; Low Back 'Spine Fusion' Surgery
Keywords: acupuncture; auricular acu-therapy; gua sha therapy; low back 'spine fusion'; post surgical pain; post surgical recovery; Pain and recovery from 'spine fusion' surgery
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual care alone (No Intervention): Subjects receive usual care alone before and after spine fusion surgery
- Active Intervention (Experimental): Acupuncture therapies, ear seeds, acupuncture treatment and gua sha, designed to reduce pain and facilitate recovery for low back spine fusion patients.
  Interventions: Procedure: Acupuncture therapies
- Control Arm (Sham Comparator): Indirect therapies with same encounter time and timing as direct care group.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Acupuncture therapies — Acupuncture therapies combined in treatment: application of ear seeds; acupuncture; and acupuncture with gua sha treatment designed to relieve pain and facilitate recovery.
  Other Names: Acupuncture auricular therapy; Acupuncture therapy; Gua sha therapy
  Arms: Active Intervention
Procedure: Control — Indirect therapies that mimic direct therapy intervention
  Other Names: Indirect auricular therapy; Indirect acupuncture therapy
  Arms: Control Arm

SUMMARY:
Acupuncture has been studied in the perioperative setting and shown to reduce pain, anxiety, nausea and vomiting. Studies have been conducted in orthopedic surgery patients, but not spine patients. The investigators study will look at a combination of acupuncture therapies for patients having low back spine fusions to assess pain levels and return to function.

114 subjects will be randomized into a direct acupuncture therapy group (38), an indirect acupuncture therapy group (38), or usual care alone (38). All subjects will receive usual care for spine fusion patients.

Direct acupuncture therapy subjects will have pre-op auricular seeds in four distinct ear points bilaterally, an acupuncture treatment on the day after surgery and an acupuncture treatment with gua sha on the 2nd day after surgery (typically day of discharge).

The indirect acupuncture therapy group will have treatment timed exactly as the direct intervention group but consist of 'indirect' treatment: tape placed at ear points at pre-op, ear seeds placed on several body points on the first and second day after surgery.

BPI, VAS, SPF36-2, and ODI measures will be taken at enrollment and at the 4-6 week follow-up appointment with subjects' spine surgeon. BPI and VAS will also be taken at day 3 and day 7-10 additionally.

DETAILED DESCRIPTION:
Active treatment will involve 3 acupuncture therapy sessions. The first encounter takes place in the holding area just prior to surgery. Subjects will have ear seeds (vacaria seeds prefixed to tape) placed on four ear points bilaterally: Shen men, Heart, Liver and Lumbar region point. These will remain on the ear for the duration of surgery and through discharge. If any one of the seeds falls off, it will be replaced at the next intervention session.

The second active session will include acupuncture needling at body points: some mandated, and some selected from listed options representing flexibility to individualize a treatment. Subject is likely in a supine position or sitting.

At third active intervention the subject will be positioned on body cushion in their hospital bed, prone. Light Gua sha will be applied at the paraspinal region above the surgical area, and across the gluteus medius area below same. If calves are tight or painful, light Gua sha may be applied. Mandated acupuncture points will be needled with selection of additional points based on pain and symptom presentation.

The control arm includes three encounters of 'indirect acupuncture therapy' timed identically to the active arm. In the first instead of ear seeds, blank pieces of tape will be applied to the subjects ears bilaterally in the holding area just prior to surgery.

The second encounter the subject will have their ear tape renewed if necessary; and 'vacaria seeded tape' will be fixed to the 'four-gates': Large Intestine 4 on the hand and Liver 3 on the foot and left in place for 20-25 minutes and then removed.

The final session will be a repeat of the second session.

Subjects will be told that the study is comparing kinds of acupuncture treatment: direct and indirect.

The third arm will be usual care alone. All subjects will receive usual care in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* English speaking
* Admitted for lumbar spine surgery

Exclusion Criteria:

* No serious psychiatric illness
* Subject has not had acupuncture for four weeks prior to surgery
* Subject agrees to not have elective acupuncture for 6 weeks after surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pain scores on Visual Analog Scale and Brief Pain Inventory | 3rd day, 7-10 days and at 4-6 weeks
  Does this combination of acupuncture therapies: ear seeds, acupuncture and acupuncture with gua sha given in hospital before and after low back 'spine fusion' surgery reduce pain over a 4-6 week period of recovery compared to control and usual care alone.

SECONDARY OUTCOMES:
Measure of 'return to function' on Short form Survey Instrument (SF-36) and Oswestry Disability Index (ODI) from baseline to '4-6 week' follow-up | 4-6 weeks
  Does this combination of acupuncture therapies: ear seeds, acupuncture and acupuncture with gua sha given in hospital before and after low back 'spine fusion' surgery facilitate return of function over a 4-6 week period of recovery compared to control and usual care alone.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Nielsen, PhD, Principal Investigator — Beth Israel Medical Center Integrative Medicine Department
Locations (1):
- Beth Israel Medical Center Orthopedic Surgery, Spine Center, New York, New York, United States